CLINICAL TRIAL: NCT00813540
Title: The Effects of Exercise Training on the Health-related Fitness of Colon Cancer Survivors: a Randomized Controlled Trial
Brief Title: The Effects of Exercise Training on the Health-related Fitness of Colon Cancer Survivors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G1-23950
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2012-04

CONDITIONS: Colonic Neoplasms
Keywords: Colonic Neoplasms; Aerobic Exercise; Weight Lifting; Body Composition
MeSH Terms: conditions — Colonic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Exercise
  Interventions: Behavioral: Exercise Training
- 2 (Other): Usual Care, no intervention
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Exercise Training — The exercise group will perform supervised stationary cycle ergometer exercise 3 times per week for 12 weeks and be progressed from 15 to 45 minutes and 60% to 110% of the power output obtained at V02peak. Resistance training will be completed twice per week and will include exercises for all major muscle groups. The training will progress from 60% to 80% of 1RM over the course of the intervention.
  Arms: 1
Other: Usual Care — Usual Care
  Arms: 2

SUMMARY:
Recent studies have suggested that individuals diagnosed with colon cancer who are inactive and/or overweight, may have poorer survival outcomes. Exercise training has been shown to improve fitness and body composition in other cancer survivor groups. The investigators hypothesize that an exercise training program will be a safe, feasible, and effective intervention to improve the fitness and body composition of a group of colon cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage II or III colon cancer diagnosis
* Less than or equal to 1 year since the completion of all adjuvant treatment
* Negative Physical Activity Readiness Questionnaire (PAR-Q) or completed Physical Activity Readiness Medical Examination (PARmed-X) form
* 18 years of age or older
* Ability to understand and provide written informed consent in English
* Willingness to be randomized
* Willingness to complete outcome measures at each assessment time point
* Available for the duration of study intervention period
* Able to travel to our fitness centre 3/week for the study period

Exclusion Criteria:

* Any absolute contraindication to to exercise testing or training
* Evidence of active disease (metastatic, recurrent, or unresectable colon cancer)
* Any uncontrolled medical condition or psychiatric illness that would prevent completion of the exercise program or interfere with the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety (Monitoring for Adverse Events) | 12 Weeks

SECONDARY OUTCOMES:
Change in Aerobic Capacity | Baseline and 12 Weeks
Change in body composition | Baseline and 12 Weeks
Feasibility (Adherence to the exercise training program) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Courneya, Ph.D., Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institue, Edmonton, Alberta, Canada